CLINICAL TRIAL: NCT03812250
Title: EUS-guided Biliary Drainage vs. ERCP Assisted Transpapillary Drainage for Malignant Biliary Obstruction: a Randomized Clinical Trial
Brief Title: EUS-guided Biliary Drainage vs. ERCP Assisted Transpapillary Drainage for Malignant Biliary Obstruction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: First People's Hospital of Hangzhou (Other)
Responsible Party: Principal Investigator, Jianfeng Yang, Hangzhou First People's Hospital, First People's Hospital of Hangzhou
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2018
Record Dates: First submitted 2019-01-15; First posted 2019-01-23 (Actual); Last update posted 2023-02-21 (Actual); Status verified 2023-02

CONDITIONS: Malignant Biliary Obstruction

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ERCP assisted trans-papillary drainage (Active Comparator): ERCP assisted trans-papillary drainage for malignant biliary obstruction
  Interventions: Procedure: ERCP assisted trans-papillary drainage for malignant biliary obstruction
- EUS-guide biliary drainage (Active Comparator): EUS-guide biliary drainage for malignant biliary obstruction
  Interventions: Procedure: EUS-guide biliary drainage for malignant biliary obstruction

INTERVENTIONS:
Procedure: ERCP assisted trans-papillary drainage for malignant biliary obstruction — ERCP assisted trans-papillary drainage for malignant biliary obstruction
  Arms: ERCP assisted trans-papillary drainage
Procedure: EUS-guide biliary drainage for malignant biliary obstruction — EUS-guide biliary drainage for malignant biliary obstruction
  Arms: EUS-guide biliary drainage

SUMMARY:
Purpose of the study: To compare efficacy, stent patency, re-intervention rate, cost, quality of life, survival time, and adverse events between EUS-guide biliary drainage (EUS-BD) and ERCP assisted trans-papillary drainage for malignant biliary obstruction.

Subjects of the study: Patients who have malignant biliary obstruction.

Methods of the study:

* Prospective randomized controlled study
* Patients were randomly divided into two groups, EUS-BD group or ERCP group
* Patients will get assigned procedure (EUS-BD or ERCP assisted trans-papillary drainage)for decompression of malignant biliary obstruction
* After the procedure, regular follow up, blood test, and imaging test will be done to check sufficient biliary decompression, stent patency, re-intervention rate, cost, quality of life, survival time, and adverse events rate.

Statistical methods: SPSS 23.0 statistical software was used. The measurement data was expressed as x± s, and t-test or non-parametric test was used. Chi-square test was used for count data.

DETAILED DESCRIPTION:
ERCP is a well-established procedure for the management of malignant biliary obstruction. However, even in expert hands, ERCP fails in 3%-5% of cases, especially in patients with surgically altered anatomy or difficult biliary cannulation. In these cases, more invasive options are usually considered, which including percutaneous trans-hepatic biliary drainage and surgical intervention, but they all have been associated with a higher risk of complications and prolonged hospital stay. EUS-guide biliary drainage using a metal stent, particularly a lumen-apposing metal stent, is a promising technique for biliary decompression in patients with failed ERCP. There has been growing global experience with EUS-BD in recent years, and data from expert centers support the feasibility and efficacy of EUS-BD. However, few researches compared the efficacy and complication rates between EUS-BD and ERCP for malignant biliary obstruction. The investigators herein aim to conduct a randomized controlled clinical trial to compare the efficacy and complication rates between EUS-BD and ERCP for malignant biliary obstruction.

ELIGIBILITY:
Inclusion Criteria:

* age: 18 - 85 years
* a patients who had malignant biliary obstruction confirmed by imaging examinations and Pathological examination
* Hyperbilirubinemia (total bilirubin >= 1.5 mg/dl)
* inoperable state
* patients who agree to join this study

Exclusion Criteria:

* a patients who cannot endure sedation or therapeutic endoscopic procedure
* a patients with bleeding tendency (PT > 1.5 INR, PLT < 50,000)
* patients underwent biliary drainage by surgery, ERCP or percutaneous transhepatic biliary drainage

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2023-02-10 (Actual); Study Completion 2023-02-15 (Actual)

PRIMARY OUTCOMES:
Clinical success rates | one month after the procedures.
  The number of patients with total bilirubin drop more than 50 % compared with baseline after successful endoscopic procedures.
Adverse events rates | within 6-9 months after the procedures
  The number of patients who developed adverse events, included biliary leakage, hemorrhage, perforation, cholangitis as defined and graded according to the consensus guideline.

SECONDARY OUTCOMES:
Re-intervention rates | within 6-9 months from the procedures
  Number of re-interventions (ERCP or PTCD) that are necessary after successful endoscopic treatment (for example due to stent migration or stent occlusion)
Evaluation of the cost of the procedure and hospitalization. | Up to 30 days after the intervention.
  Evaluation of the cost for different procedures.
overall survival | within 6-9 months from the procedures
  death in the follow up after endoscopic treatment

CONTACTS AND LOCATIONS:
Overall Officials: Xiaofeng Zhang, M.D., Principal Investigator — First People's Hospital of Hangzhou
Locations (1):
- Hangzhou First People's Hospital, Hangzhou, China

REFERENCES:
- [Result] Park JK, Woo YS, Noh DH, Yang JI, Bae SY, Yun HS, Lee JK, Lee KT, Lee KH. Efficacy of EUS-guided and ERCP-guided biliary drainage for malignant biliary obstruction: prospective randomized controlled study. Gastrointest Endosc. 2018 Aug;88(2):277-282. doi: 10.1016/j.gie.2018.03.015. Epub 2018 Mar 30. PMID 29605722